CLINICAL TRIAL: NCT01030237
Title: An Evaluation of the Safety and Efficacy of FID 114657
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-07-34
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114657 (Experimental): FID 114657
  Interventions: Other: FID 114657
- Soothe XP Lubricant Eye Drops (Active Comparator): Soothe XP Lubricant Eye Drops
  Interventions: Other: Soothe XP Lubricant Eye Drops

INTERVENTIONS:
Other: FID 114657 — 1 drop both eyes four times a day for 6 weeks
  Arms: FID 114657
Other: Soothe XP Lubricant Eye Drops — 1 drop both eyes four times a day for 6 weeks
  Arms: Soothe XP Lubricant Eye Drops

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of FID 114657 in comparison to Soothe XP in a specified population of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye
* NaFl Corneal Staining sum score ≥ 3 in either eye

Exclusion Criteria:

* Must not have worn contact lenses for 1 week preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Tear Break-Up Time (TBUT) | measured at Days 0, 7, 14, 28 and 42
Corneal Staining | measured at Days 0, 7, 14, 28 and 42
Conjunctival Staining | measured at Days 0, 7, 14, 28 and 42